CLINICAL TRIAL: NCT03070756
Title: Extended Evaluation of the Efficacy of a Proactive FOT-based Auto-CPAP Algorithm in Patients With Predominantly Obstructive Sleep Apnea
Brief Title: Extended Evaluation of the Efficacy of a Proactive FOT-based Auto-CPAP Algorithm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heinen und Löwenstein GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Organization: Heinen (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-pLINE-AC-1
Record Dates: First submitted 2016-08-09; First posted 2017-03-06 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: auto-CPAP; forced oscillation technique; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment group (auto-CPAP) (Other): Participants of this study undergo an diagnostic PSG night. The diagnostic night is followed by an auto-CPAP treatment night.
  Interventions:
  The treatment night is in line with the routine procedure of the laboratory except the following intervention: the device settings for the treatment night are applied according to the study protocol (minimal intervention).
  Interventions: Device: Minimal-Intervention - Specification of device settings

INTERVENTIONS:
Device: Minimal-Intervention - Specification of device settings — - device settings for auto-CPAP treatment night: therapy mode=APAP, Pmin=5hPa,Pmax=20 hPa, Soft-Start duration <=15 min, softPAP Level is selected based on patient comfort
  Other Names: Specification of device settings

SUMMARY:
This study implements an extended (post marked) examination of the efficacy of a proactive auto-CPAP algorithm, which is based on the forced oscillation technique (FOT) in a sample of patients with predominantly obstructive sleep apnea. The auto-CPAP algorithm examined in this study is implemented in the medical devices prisma20A and prismaLAB (Löwenstein Medical Technology).

DETAILED DESCRIPTION:
Patients diagnosed with obstructive sleep apnea and who comply with inclusion criteria of the study will be informed about the possibility of participation. Following informed and written consent, participants will undergo a PSG-diagnostic night according to clinical routine, followed by an auto-CPAP treatment night with a prismaLINE device (prismaLAB or prisma20A). The device settings applied in the treatment night are defined by the study protocol (see interventions). Following the auto-CPAP treatment night, study participation is completed. Any following treatment and patient care is administered according to clinical routine.

Primary and secondary outcome measures of sleep stage and respiratory event indices are evaluated at diagnostic night and auto-CPAP treatment night.

The enrollment consists of two phases. During phase 1 (training phase) 10 participants are enrolled and complete the study protocol. Phase 1 serves as a training phase to establish a common standard of data quality and acquisition. Data of the training phase are not included in the statistical analysis. Following the training phase the efficacy of the auto-CPAP algorithm is evaluated in a sample of 70 participants.

ELIGIBILITY:
Inclusion Criteria:

* Apnea-Hypopnea Index (AHI) > 15,0 (n/h Total Sleep Time)
* Initial diagnosis of predominant obstructive sleep apnea (percentage of central respiratory events < 20 %)
* informed written consent

Exclusion Criteria:

* missing informed written consent
* Participation in another clinical trial that influences the initiation of auto-CPAP treatment by specifications of device settings or titration procedure
* acute cardiac decompensation
* severe arrhythmia
* severe hypotension, particularly in combination with intravascular volume depletion
* severe epistaxis
* high risk of barotrauma
* decompensated pulmonary conditions
* pneumothorax or pneumomediastinum
* pneumocephalus
* cranial trauma
* status following brain surgery or surgical intervention on the pituitary gland or the middle/inner ear
* acute sinus infection (sinusitis), middle ear infection (otitis media) or perforated eardrum
* dehydration

Exclusion Criteria Statistical Evaluation:

Data of patients who completed the study protocol will be excluded from statistical analysis if one of the following criteria applies:

* non adherence to in-/exclusion criteria
* AHI <= 15,0 (n/h TST) or percentage of central respiratory events >= 20% in the second, study specific PSG-diagnostic night
* application of incorrect device settings
* insufficient data quality of PSG-acquisition
* the device was applied outside range of indication
* data of diagnostic night are not acquired as a PSG
* total time of softSTART duration exceeded 60 min
* the auto-CPAP device was restarted >= 3 times during the treatment night. Recurrent reductions of device therapy pressure to start level (device restarts) which are applied within a time frame of <= 5 minutes after another restart will be assigned to previous restart und therefore numbered as one. Restarts which take place before initial falling asleep will not be numbered.
* the application time of the auto-CPAP device was <6h during treatment night

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI /h TST) | 2 days: change from recorded AHI in diagnostic PSG-acquistion to recorded AHI in treatment PSG-acquistion
  number of apneas and hypopneas per hour of sleep time (TST)

SECONDARY OUTCOMES:
Obstructive Apnea-Hypopnea Index (oAHI /h TST) | 2 days: diagnostic and treatment PSG-acquistion
  number of obstructive apneas and hypopneas per hour of sleep time (TST)
Obstructive Apnea Index (oAI /h TST) | 2 days: diagnostic and treatment PSG-acquistion
  number of obstructive apneas per hour of sleep time (TST)
Central Apnea-Hypopnea Index (cAHI /h TST) | 2 days: diagnostic and treatment PSG-acquistion
  number of central apneas and hypopneas per hour of sleep time (TST)
Oxygen Desaturation Index (ODI /h TST) | 2 days: diagnostic and treatment PSG-acquistion
  number of oxygen desaturations per hour of sleep time (TST)
Arousal Index (ArI /h TST) | 2 days: diagnostic and treatment PSG-acquistion
  number of arousals per hour of sleep time (TST)
Respiratory Arousal Index (ArI_resp /h TST) | 2 days: diagnostic and treatment PSG-acquistion
  number of respiratory arousals per hour of sleep time (TST)
Snore (Snore /% TST) | 2 days: diagnostic and treatment PSG-acquistion
  Percentage of total sleep time with snoring
Slow-wave sleep (N3 /% TST) | 2 days: diagnostic and treatment PSG-acquistion
  Percentage of total sleep time with slow wave sleep
therapy pressure /hPa | 1 day: treatment night (auto-CPAP)
  P95, P90 and median treatment pressure (hPa) in auto-CPAP night with prismaLINE
leakage / l/min | 1 day: treatment night (auto-CPAP)
  P95, percentage of therapy time with leakage > 50 l/min and median leakage during auto-CPAP treatment night.
Time in Bed with oxygen saturation < 90% (SpO2 < 90 % / %TIB) | 2 days: diagnostic and treatment PSG-acquistion
  Percentage of time in Bed with an oxygen sturation < 90 %

CONTACTS AND LOCATIONS:
Overall Officials: Winfried J. Randerath, Professor, Study Director — Wissenschaftliches Institut Bethanien e.V
Locations (1):
- Wissenschaftliches Institut Bethanien e.V., Solingen, Germany

IPD SHARING:
Plan to Share IPD: No